CLINICAL TRIAL: NCT02204371
Title: A Phase II Study to Evaluate the Effects of up to 12 Weeks of Pazopanib Dosing on Bleeding in Subjects With Hereditary Haemorrhagic Telangiectasia
Brief Title: Evaluation of Pazopanib on Bleeding in Subjects With Hereditary Haemorrhagic Telangiectasia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated as the asset was sold to another company who decided not to pursue this indication with this drug.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201128
Record Dates: First submitted 2014-07-28; First posted 2014-07-30 (Estimated); Results first posted 2017-07-06 (Actual); Last update posted 2017-07-06 (Actual); Status verified 2017-04

CONDITIONS: Telangiectasia, Hereditary Hemorrhagic
Keywords: Pazopanib; hereditary haemorrhagic telangiectasia; bleeding
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic; Hemorrhage | interventions — pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part A- Dose Escalation phase (Experimental): Part A will be an open label, dose-escalation study in which 4 cohorts of approximately 6 subjects will receive increasing doses of pazopanib for a maximum of 12 weeks. The dose in the first cohort will be 50mg per day and the maximum dose in a cohort will be 400 mg per day. Dose escalation will not occur if the predefined safety stopping criteria are met or at least 4 subjects in a cohort have demonstrated efficacy. Cohort 4 receiving 400 mg dosing schedule may involve cycles of up to 3 weeks of active treatment, followed by up to 3 weeks wash-out (instead of 12 weeks continuous dosing). Decision will be based on safety data obtained from lower doses
  Interventions: Drug: Pazopanib
- Part B-Dose Optimization phase (Experimental): If efficacy is demonstrated in Part A with an acceptable safety profile, Part B will be initiated to further define the optimal dose(s) including dose duration/schedule and to provide further support for the proof of mechanism. Approximately 15 subjects will participate and will be randomised to active or placebo in a ratio of 3:2. This part of the study will be double-blind
  Interventions: Drug: Pazopanib; Drug: Placebo

INTERVENTIONS:
Drug: Pazopanib — Pazopanib is available as 50 mg and 200 mg tablets to be administered orally once daily in the morning at least one hour before or two hours after a meal for 12 weeks
Drug: Placebo — Pazopanib matching placebo is available as tablets to be administered orally once daily in the morning at least one hour before or two hours after a meal for 12 weeks
  Arms: Part B-Dose Optimization phase

SUMMARY:
This study will investigate whether pazopanib can reduce epistaxis and improve anaemia in subjects with hereditary haemorrhagic telangiectasia (HHT) at a dose that is well tolerated. The study will have 2 parts. Part A will be an open label, dose-escalation study in which up to 4 cohorts of approximately 6 subjects each will receive increasing doses of pazopanib for a maximum of 12 weeks. The dose in the first cohort will be 50mg per day and the maximum dose in a cohort will be 400 mg per day. Dose escalation will not occur as planned if the predefined safety stopping criteria are met or at least 4 subjects in a cohort have demonstrated efficacy (as measured by epistaxis, haemoglobin, transfusion or iron infusion requirements). If efficacy is demonstrated in Part A with an acceptable safety profile, Part B will be initiated to further define the optimal dose(s) including dose duration/schedule and to provide further support for the proof of mechanism. Approximately 15 subjects will participate and will be randomised to active or placebo in a ratio of 3:2. This part of the study will be double-blind.

ELIGIBILITY:
Inclusion Criteria:

* Males/females aged between 18 and 75 years of age inclusive, at the time of signing the informed consent.
* Diagnosis of definite or possible HHT by the Curaçao criteria. According to the Curaçao criteria, a definite diagnosis of HHT is defined as having at least 3 of the following criteria while a possible diagnosis is defined as 2 criteria: a) spontaneous and recurrent epistaxis; b) multiple telangiectasias at characteristic sites: lips, oral cavity, fingers, nose; c) visceral lesions: gastrointestinal (GI) telangiectasia, pulmonary, hepatic, cerebral or spinal arteriovenous malformations (AVMs); d) a first degree relative with HHT according to these criteria.
* Subject meets at least one of the following criteria: a) Severe epistaxis over previous 4 weeks defined as an average of at least 3 nose bleeds per week AND a total duration of greater than 15 min per week AND requiring iron therapy (oral and/or intravenous); b) Moderate or severe iron deficiency anaemia (Hgb < 11gram [g]/deciliter [dL], at screening) despite iron infusions (at least 0.5g iron per month) or blood transfusions (at least 2 units per month) AND substantial compromise in the quality of life according to the investigator (e.g. nose bleeds, lethargic, cannot maintain job, listless, fatigue). Anaemia must be HHT related in the opinion of the investigator, ie: due to HHT-defined bleeding (epistaxis and/or bleeding from the GI tract [presence of telangiectatic lesions, exclusion of active ulcer disease or other infection, inflammation]), and lack of other known etiologies such as blood dyscrasias.
* Epistaxis (if applicable) is considered to be clinically stable during the 4 weeks prior to Screening in the clinical judgment of the investigator (i.e. no major changes in frequency or duration of epistaxis).
* A female subject is eligible to participate if she is of non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy [for this definition, "documented" refers to the outcome of the investigator's/designee's review of the subject's medical history for study eligibility, as obtained via a verbal interview with the subject or from the subject's medical records]; or postmenopausal defined as 12 months of spontaneous amenorrhoea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 milli-international units per milliliter (MIU/mL) and estradiol < 40 picogram per milliliter (pg/mL) (<147 picomole per liter [pmol/L]) is confirmatory].
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Subject is able and willing to return for outpatient visits at the protocol specified intervals.
* Subject agrees not to undergo laser ablation of nasal telangiectasias or take any experimental therapies for HHT other than the study drug while participating in the study (over the counter medications, topical treatments, nasal hygiene and palliative therapies are acceptable as long as use is consistent). If subjects stop taking experimental therapies on entry to the study there should be a wash-out period of at least 5 half-lives prior to the start of the run-in).
* Based on averaged corrected QT either Bazett's formula (QTcB), Fridericia's formula (QTcF) values of triplicate ECGs obtained over a brief recording period: QTc < 450 milliseconds (msec); or QTc < 480 msec in subjects with Bundle Branch Block.

Exclusion Criteria:

* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones; and with the exception of vascular abnormalities that are related to the HHT).
* Subject has known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to pazopanib that in the opinion of the investigator contradicts their participation.
* Currently has untreated cerebral vascular malformations (CVMs) (Note: magnetic resonance imaging [MRI] scan does not need to be repeated at Screen if CVMs were absent on scan after age 18 years or in the last 5 years).
* Currently has known pulmonary AVMs with feeding artery diameter >3 millimeter (mm).
* Symptomatic liver AVMs (defined as chronic right upper quadrant pain, symptomatic portal hypertension or heart failure).
* Known significant bleeding sources other than nasal or gastrointestinal.
* Systemic use of a vascular endothelial growth factor (VEGF) inhibitor in the past 12 weeks or previous enrolment in this study.
* Current use of anticoagulants including but not limited to vitamin K antagonists (e.g., warfarin) at any dose; unfractionated or low molecular weight heparins at standard doses for treatment of venous thromboembolism (VTE) (e.g., enoxoparin); antiplatelets (e.g., clopidogrel), or direct factor Xa inhibitors (e.g., apixaban). Use of low dose aspirin <= 81mg is allowed as long as use is consistent.
* Active and recent onset diarrhoea.
* Current or recent malignancies (except non-melanoma skin cancers) Subject has: a) had major surgery (eg, surgical ligation of an AVM) or trauma within 28 days; b) had minor surgical procedures (eg, central venous access line removal) within 7 days prior to dosing; c) any non-healing wound, fracture or ulcer
* Subject has clinically significant gastrointestinal abnormalities (other than HHT-related vascular lesions) including, but not limited to: malabsorption syndrome, major resection of the stomach or small bowel that could affect the absorption of study drug (eg, short bowel syndrome), active peptic ulcer, known intraluminal metastatic lesions/s with suspected bleeding, inflammatory bowel disease, ulcerative colitis or other gastrointestinal conditions with increased risk of perforation, lifetime history of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess
* Subject has a history of cerebrovascular accident (including transient ischaemic attacks), pulmonary embolism or untreated deep vein thrombosis (DVT) within the 6 months prior to first dose of study drug.
* Subject has a history of any one or more of the following cardiovascular conditions within the 6 months prior to first dose of study drug: cardiac angioplasty or stenting, myocardial infarction, unstable angina, ischaemic stroke, symptomatic peripheral vascular disease
* Class III or IV congestive heart failure, as defined by the New York Heart Association (NYHA).
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* Hgb < 7 gram per deciliter (g/dL).
* Platelets < 100x10^9/L, International normalized ratio (INR) > 1.2x upper limit of normal (ULN) and activated partial thromboplastin time (aPTT) >1.2xULN.
* Alanine aminotransferese (ALT) >= 2xULN or bilirubin > 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).

Subject has poorly controlled hypertension [defined as systolic blood pressure (SBP) >= 140 millimeter of mercury (mmHg) or diastolic blood pressure (DBP) >= 90mmHg]. Initiation or adjustment of antihypertensive medication(s) is permitted prior to study entry. At Screening, blood pressure must be assessed three times and the mean SBP/DBP must be <140/90 mmHg in order for a subject to be eligible for the study.

* Substantive renal disease (estimated glomerular filtration rate [eGFR] < 60 mL/minute/1.73 meter^3 calculated using the Cockcroft-Gault formula)
* Thyroid stimulating hormone > ULN.
* Urine protein creatinine ratio >0.3
* White blood cell count< 3500/mm^3.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the start of the run-in period: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Unable or unwilling to discontinue use of prohibited medications mentioned below for at least 14 days or 5 half-lives of a drug (whichever is longer) prior to the start of the run-in period and for the duration of the study. Medications that inhibit Cytochrome P450 3A4 (CYP3A4) may result in increased plasma pazopanib concentrations; therefore, co-administration of strong CYP3A4 inhibitors is PROHIBITED beginning 14 days prior to the first dose of study treatment until 15 days after the last dose of pazopanib. Strong CYP3A4 inhibitors include (but are not limited to): Antibiotics: clarithromycin, telithromycin, troleandomycin; human immunodeficiency virus (HIV): protease inhibitors (ritonavir, indinavir, saquinavir, nelfinavir, amprenavir, lopinavir); Antifungals: itraconzaole, ketoconazole, voriconazole, fluconazole; Antidepressants: nefazodone, Miscellaneous: grapefruit, grapefruit juice or other grapefruit product. statins, anticoagulants and tamoxifen use is prohibited.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2015-02-25 (Actual); Primary Completion 2016-02-10 (Actual); Study Completion 2016-02-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (6):
- United States (5):
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Augusta, Georgia
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Salt Lake City, Utah
- GSK Investigational Site, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was planned as a two part study (Part A and Part B). As efficacy based dose escalation stopping criteria was met, there was only one dose cohort (50 milligrams [mg] once daily cohort) in Part A. The study was stopped prior to Part B being conducted.
Pre-assignment Details: Run-in period started at the screening visit or up to 2 weeks after the screening visit. Participants (par.) were stabilized on a anemia management plan for 4-8 weeks prior to the first dose. Unstable par. were allowed to continue in the run-in period for additional 4 weeks. 2 par. did not met the eligibility criteria.
Groups:
- GW786034 50 mg Once Daily: Participants with hereditary hemorrhagic telangiectasia (HHT) received GW786034 50 mg tablet orally once daily at least one hour before or two hours after a meal in the morning for up to 12 weeks in the open label non-randomized phase.
Period: Overall Study
Arm/Group | GW786034 50 mg Once Daily
Started | 7
Completed | 6
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | GW786034 50 mg Once Daily
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.3 (9.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 3
Race/Ethnicity, Customized [Number; unit: Participants]
  White - White/Caucasian/European Heritage | 7

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Epistaxis Severity Score at the Indicated Time Points
Description: The Epistaxis (nose bleeding) severity score (ESS) is a 6-item par-reported outcome measure designed to be a uniform epistaxis severity scoring system to assess the effectiveness of specific treatments on HHT-related epistaxis. Four questions document epistaxis frequency, duration, intensity and need for treatment, whereas two additional questions detail the presence of anemia and if a par has required a blood transfusion as a consequence of their epistaxis. Questions are variably weighted and results are tabulated on a 0-10 scale (0=no disease, 10 = severe disease). The minimum important difference is 0.71. Baseline is the Day1 pre-dose assessment value. Change from Baseline is calculated as the Post dose value at the indicated visit minus the Baseline value. Par were evaluated at Baseline, Treatment period (Weeks 6 and 12) and Follow-up period (Weeks 16, 20, 24 and 28). Only those par available at the indicated timepoints were analysed (specified by n=X in the category titles).
Time Frame: Baseline, Week 6, Week 12, Week 16, Week 20, Week 24 and Week 28
Population: Pharmacodynamic Population: All par. who received at least one dose of study treatment (Safety Population) and who also provided data from at least one pharmacodynamic assessment (hemoglobin, ferritin, epistaxis daily diary).
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | GW786034 50 mg Once Daily
Number analyzed (Participants) | 7
Scores on a scale
  Week 6, n=7 | -0.59 (0.802)
  Week 12, n=6 | -1.16 (1.023)
  Follow-up Week 16, n=7 | -0.60 (1.299)
  Follow-up Week 20, n=6 | -1.41 (1.674)
  Follow-up Week 24, n=5 | -1.27 (1.519)
  Follow-up Week 28, n=5 | -0.08 (1.920)

2. Primary Outcome: Change From Baseline in the Average of the Last 3 Hemoglobin Measures in the Dosing Period (Week 9, Week 10.5 and Week 12)
Description: For post-Baseline hemoglobin assessments, average of the last 3 measurements of the dosing period (Weeks 9, 10.5 and 12) was computed. Only pre-transfusion hemoglobin values have been included in the analyses. Baseline hemoglobin value is the average of the last two measurements during the run-in period. . Average of the last two measurements during the run-in period was calculated as sum of the last 2 measured values of hemoglobin divided by 2. Change from Baseline was calculated as the average of the last 3 measured values of hemoglobin minus the Baseline value. Average of the last 3 measurements was calculated as sum of the last 3 measured values of hemoglobin divided by 3. If measurements were missing at one or two of the 3 visits at Weeks 9, 10.5 and 12, then the average was based on the available measurements.
Time Frame: Baseline, Week 9, Week 10.5 and Week 12
Population: Pharmacodynamic Population. Only those par. available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Grams per liter (g/L)
Arm/Group | GW786034 50 mg Once Daily
Number analyzed (Participants) | 6
Grams per liter (g/L) | 7.58 (17.543)

3. Primary Outcome: Change From Baseline in Hemoglobin at the Indicated Time Points
Description: Only pre-transfusion hemoglobin values have been included in the analyses. All hemoglobin values that fall within 5 days of packed red blood cells (PRBC) transfusion are considered as post-transfusion values. Baseline hemoglobin value is defined as the average of the last two measurements during the run-in period. Average of the last two measurements during the run-in period was calculated as sum of the last 2 measured values of hemoglobin divided by 2. Change from Baseline was calculated as the Post dose value at the indicated visit minus the Baseline value. Par. were evaluated at Treatment period (Weeks 1.5, 3, 4.5, 6, 7.5, 9, 10.5 and 12) and Follow-up period (Weeks 16, 20, 24 and 28).
Time Frame: Baseline, Week 1.5, Week 3, Week 4.5, Week 6, Week 7.5, Week 9, Week 10.5, Week 12, Week 16, Week 20, Week 24 and Week 28
Population: Pharmacodynamic Population. Only those par. available at the indicated time points were analyzed (specified by n=X in the category titles).
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | GW786034 50 mg Once Daily
Number analyzed (Participants) | 7
g/L
  Week 1.5, n=7 | 7.50 (11.113)
  Week 3, n=6 | 11.92 (13.492)
  Week 4.5, n=7 | 7.50 (22.042)
  Week 6, n=7 | 6.48 (19.967)
  Week 7.5, n=6 | 8.83 (12.770)
  Week 9, n=6 | 6.67 (14.865)
  Week 10.5, n=6 | 7.50 (15.485)
  Week 12, n=6 | 8.58 (25.150)
  Follow-Up Week 16, n=7 | 7.00 (22.739)
  Follow-Up Week 20, n=6 | 7.56 (19.212)
  Follow-Up Week 24, n=5 | 4.93 (11.086)
  Follow-Up Week 28, n=5 | -3.80 (7.926)

4. Primary Outcome: Duration of Epistaxis Over the Last 2 Weeks of the Dosing Period and by Time Over the Entire Dosing and Follow-up Period by 2 Week Interval (From Daily Diaries)
Description: Duration of epistaxis based on daily diaries has been reported over Baseline, On-Therapy (OT) to Follow-up (F). Individual participant data from the daily diaries has been reported.
Time Frame: Over last 2 weeks of the run-in phase and then 2 week intervals throughout treatment period and follow-up period (from daily diaries)
Population: Pharmacodynamic Population
Measure: Number; unit: Minutes
Arm/Group | GW786034 50 mg Once Daily
Number analyzed (Participants) | 7
Minutes
  Participant 1, Baseline | 26
  Participant 1, OT Day1-13 | 28
  Participant 1, OT Day 14-27 | 32
  Participant 1, OT Day 28-41 | 32
  Participant 1, OT Day 42-55 | 34
  Participant 1, OT Day 56-69 | 26
  Participant 1, OT Day 70 - 83 | 30
  Participant 1, F Day 1-14 | 22
  Participant 1, F Day 15 - 28 | 28
  Participant 1, F Day 29 - 42 | 34
  Participant 1, F Day 43 - 56 | 43
  Participant 1, F Day 57 - 70 | 33
  Participant 1, F Day 71 - 84 | 27
  Participant 1, F Day 85 - 98 | 46
  Participant 1, F Day 99 - 112 | 66
  Participant 2, Baseline | 846
  Participant 2, OT Day1-5 | 301
  Participant 2, OT Day 6 - 19 | 966
  Participant 2, OT Day 20 - 33 | 1288
  Participant 2, OT Day 34 - 47 | 980
  Participant 2, OT Day 48 - 61 | 589
  Participant 2, OT Day 62 - 75 | 594
  Participant 2, OT Day 76 - 89 | 386
  Participant 2, F Day 1 - 14 | 240
  Participant 2, F Day 15 - 28 | 191
  Participant 2, F Day 29 - 42 | 426
  Participant 2, F Day 43 - 56 | 261
  Participant 2, F Day 57 - 70 | 236
  Participant 2, F Day 71 - 84 | 115
  Participant 2, F Day 85 - 98 | 467
  Participant 2, F Day 99 | 14
  Participant 3, Baseline | 130
  Participant 3, OT Day1 - 14 | 210
  Participant 3, OT Day 15 - 28 | 132
  Participant 3, OT Day 29 - 42 | 118
  Participant 3, OT Day 43 - 56 | 84
  Participant 3, OT Day57 - 70 | 65
  Participant 3, OT Day71 - 84 | 68
  Participant , F Day 1 - 14 | 127
  Participant 3, F Day 15 - 28 | 8
  Participant 3, F Day 29 - 42 | 48
  Participant 3, F Day 43 - 56 | 63
  Participant 3, F Day 57 - 70 | 70
  Participant 3, F Day 71 - 84 | 36
  Participant 3, F Day 85 - 98 | 51
  Participant 3, F Day 99 - 112 | 46
  Participant 3, F Day 113 - 115 | 5
  Participant 4, Baseline | 269
  Participant 4, OT Day1 | 30
  Participant 4, OT Day 2 - 15 | 312
  Participant 4, OT Day 16 - 29 | 125
  Participant 4, OT Day 30 - 43 | 122
  Participant 4, OT Day 44 - 57 | 93
  Participant 4, OT Day 58 - 71 | 40
  Participant 4, OT Day 72 - 85 | 40
  Participant 4, F Day 1-14 | 55
  Participant 4, F Day 15 - 28 | 84
  Participant 4, F Day 29 - 42 | 232
  Participant 4, F Day 43 - 56 | 95
  Participant 4, F Day 57 - 70 | 140
  Participant 4, F Day 71 - 84 | 79
  Participant 4, F Day 85 - 98 | 104
  Participant 4, F Day 99 - 112 | 165
  Participant 4, F Day 113 - 120 | 127
  Participant 5, Baseline | 361
  Participant 5, OT Day 1 - 2 | 63
  Participant 5 OT Day 3 - 16 | 378
  Participant 5, OT Day 17 - 30 | 404
  Participant 5, OT Day 31 - 44 | 396
  Participant 5, OT Day 45 - 58 | 211
  Participant 5, OT Day 59 - 72 | 278
  Participant 5, OT Day 73 - 86 | 202
  Participant 5, F Day 1-14 | 224
  Participant 5, F Day 15 - 28 | 130
  Participant 5, F Day 29 - 42 | 163
  Participant 5, F Day 43 - 56 | 151
  Participant 5, F Day 57 - 70 | 207
  Participant 5, F Day 71 - 84 | 170
  Participant 5, F Day 85 - 98 | 176
  Participant 5, F Day 99 - 112 | 253
  Participant 5, F Day 113 - 118 | 94
  Participant 6, Baseline | 26
  Participant 6, OT Day 1 | 0
  Participant 6, OT Day 2 - 15 | 12
  Participant 6, OT Day 16 - 29 | 28
  Participant 6, OT Day 30 - 43 | 19
  Participant 6, F Day 1-14 | 19
  Participant 6, F Day 15 - 28 | 15
  Participant 6, F Day 29 - 42 | 8
  Participant 6, F Day 43 - 56 | 26
  Participant 7, Baseline | 213
  Participant 7, OT Day 1 - 14 | 190
  Participant 7, OT Day 15 - 28 | 58
  Participant 7, OT Day 29 - 42 | 110
  Participant 7, OT Day 43 - 56 | 15
  Participant 7, OT Day 57 - 70 | 36
  Participant 7, OT Day 71 - 84 | 53
  Participant 7, F Day 1-14 | 40
  Participant 7, F Day 15 - 28 | 114
  Participant 7, F Day 29 - 42 | 68
  Participant 7, F Day 43 - 54 | 87

5. Primary Outcome: Frequency of Epistaxis Over the Last 2 Weeks of the Dosing Period and by Time Over the Entire Dosing and Follow-up Period by 2 Week Interval (From Daily Diaries)
Description: Frequency of epistaxis based on daily diaries has been reported over Baseline, On-Therapy (OT) to Follow-up (F). Individual participant data from the daily diaries has been reported.
Time Frame: as for outcome 4
Population: Pharmacodynamic Population
Measure: Number; unit: Number of nosebleeds
Arm/Group | GW786034 50 mg Once Daily
Number analyzed (Participants) | 7
Number of nosebleeds
  Participant 1, Baseline | 21
  Participant 1, OT Day1-13 | 23
  Participant 1, OT Day 14-27 | 23
  Participant 1, OT Day 28-41 | 22
  Participant 1, OT Day 42-55 | 23
  Participant 1, OT Day 56-69 | 20
  Participant 1, OT Day 70 - 83 | 25
  Participant 1, F Day 1-14 | 23
  Participant 1, F Day 15 - 28 | 24
  Participant 1, F Day 29 - 42 | 28
  Participant 1, F Day 43 - 56 | 30
  Participant 1, F Day 57 - 70 | 21
  Participant 1, F Day 71 - 84 | 23
  Participant 1, F Day 85 - 98 | 31
  Participant 1, F Day 99 - 112 | 34
  Participant 2, Baseline | 42
  Participant 2, OT Day1-5 | 17
  Participant 2, OT Day 6 - 19 | 42
  Participant 2, OT Day 20 - 33 | 55
  Participant 2, OT Day 34 - 47 | 44
  Participant 2, OT Day 48 - 61 | 32
  Participant 2, OT Day 62 - 75 | 42
  Participant 2, OT Day 76 - 89 | 37
  Participant 2, F Day 1 - 14 | 32
  Participant 2, F Day 15 - 28 | 21
  Participant 2, F Day 29 - 42 | 28
  Participant 2, F Day 43 - 56 | 28
  Participant 2, F Day 57 - 70 | 33
  Participant 2, F Day 71 - 84 | 28
  Participant 2, F Day 85 - 98 | 34
  Participant 2, F Day 99 | 3
  Participant 3, Baseline | 11
  Participant 3, OT Day1 - 14 | 17
  Participant 3, OT Day 15 - 28 | 16
  Participant 3, OT Day 29 - 42 | 13
  Participant 3, OT Day 43 - 56 | 11
  Participant 3, OT Day57 - 70 | 8
  Participant 3, OT Day71 - 84 | 13
  Participant , F Day 1 - 14 | 12
  Participant 3, F Day 15 - 28 | 3
  Participant 3, F Day 29 - 42 | 8
  Participant 3, F Day 43 - 56 | 11
  Participant 3, F Day 57 - 70 | 11
  Participant 3, F Day 71 - 84 | 5
  Participant 3, F Day 85 - 98 | 5
  Participant 3, F Day 99 - 112 | 9
  Participant 3, F Day 113 - 115 | 2
  Participant 4, Baseline | 27
  Participant 4, OT Day1 | 1
  Participant 4, OT Day 2 - 15 | 28
  Participant 4, OT Day 16 - 29 | 18
  Participant 4, OT Day 30 - 43 | 19
  Participant 4, OT Day 44 - 57 | 17
  Participant 4, OT Day 58 - 71 | 7
  Participant 4, OT Day 72 - 85 | 6
  Participant 4, F Day 1-14 | 6
  Participant 4, F Day 15 - 28 | 9
  Participant 4, F Day 29 - 42 | 18
  Participant 4, F Day 43 - 56 | 12
  Participant 4, F Day 57 - 70 | 19
  Participant 4, F Day 71 - 84 | 11
  Participant 4, F Day 85 - 98 | 12
  Participant 4, F Day 99 - 112 | 14
  Participant 4, F Day 113 - 120 | 10
  Participant 5, Baseline | 35
  Participant 5, OT Day 1 - 2 | 6
  Participant 5 OT Day 3 - 16 | 33
  Participant 5, OT Day 17 - 30 | 37
  Participant 5, OT Day 31 - 44 | 34
  Participant 5, OT Day 45 - 58 | 28
  Participant 5, OT Day 59 - 72 | 34
  Participant 5, OT Day 73 - 86 | 30
  Participant 5, F Day 1-14 | 30
  Participant 5, F Day 15 - 28 | 19
  Participant 5, F Day 29 - 42 | 22
  Participant 5, F Day 43 - 56 | 23
  Participant 5, F Day 57 - 70 | 28
  Participant 5, F Day 71 - 84 | 25
  Participant 5, F Day 85 - 98 | 27
  Participant 5, F Day 99 - 112 | 31
  Participant 5, F Day 113 - 118 | 9
  Participant 6, Baseline | 18
  Participant 6, OT Day 1 | 0
  Participant 6, OT Day 2 - 15 | 13
  Participant 6, OT Day 16 - 29 | 28
  Participant 6, OT Day 30 - 43 | 19
  Participant 6, F Day 1-14 | 17
  Participant 6, F Day 15 - 28 | 13
  Participant 6, F Day 29 - 42 | 9
  Participant 6, F Day 43 - 56 | 17
  Participant 7, Baseline | 13
  Participant 7, OT Day 1 - 14 | 9
  Participant 7, OT Day 15 - 28 | 5
  Participant 7, OT Day 29 - 42 | 11
  Participant 7, OT Day 43 - 56 | 5
  Participant 7, OT Day 57 - 70 | 5
  Participant 7, OT Day 71 - 84 | 6
  Participant 7, F Day 1-14 | 7
  Participant 7, F Day 15 - 28 | 12
  Participant 7, F Day 29 - 42 | 7
  Participant 7, F Day 43 - 54 | 6

6. Primary Outcome: Intensity of Epistaxis Over the Last 2 Weeks of the Dosing Period and by Time Over the Entire Dosing and Follow-up Period by 2 Week Interval (From Daily Diaries)
Description: Intensity of epistaxis based on daily diaries has been reported as total gushing and total non gushing from Baseline, On-Therapy (OT) to Follow-up (F). Individual participant data from the daily diaries has been reported.
Time Frame: as for outcome 4
Population: Pharmacodynamic Population
Measure: Number; unit: Number of gushing/non-gushing nosebleeds
Arm/Group | GW786034 50 mg Once Daily
Number analyzed (Participants) | 7
Number of gushing/non-gushing nosebleeds
  Participant 1, Baseline, Total Gushing | 2
  Participant 1, Baseline, Total Non-Gushing | 19
  Participant 1, OT Day1-13, Total Gushing | 0
  Participant 1, OT Day1-13, Total Non-Gushing | 23
  Participant 1, OT Day 14-27, Total Gushing | 3
  Participant 1, OT Day 14-27, Total Non-Gushing | 20
  Participant 1, OT Day 28-41, Total Gushing | 4
  Participant 1, OT Day 28-41, Total Non-Gushing | 18
  Participant 1, OT Day 42-55, Total Gushing | 3
  Participant 1, OT Day 42-55, Total Non-Gushing | 20
  Participant 1, OT Day 56-69, Total Gushing | 2
  Participant 1, OT Day 56-69, Total Non-Gushing | 18
  Participant 1, OT Day 70 - 83, Total Gushing | 2
  Participant 1, OT Day 70 - 83, Total Non-Gushing | 23
  Participant 1, F Day 1-14, Total Gushing | 0
  Participant 1, F Day 1-14, Total Non-Gushing | 23
  Participant 1, F Day 15 - 28, Total Gushing | 2
  Participant 1, F Day 15 - 28, Total Non-Gushing | 22
  Participant 1, F Day 29 - 42 , Total Gushing | 0
  Participant 1, F Day 29 - 42 , Total Non-Gushing | 28
  Participant 1, F Day 43 - 56, Total Gushing | 5
  Participant 1, F Day 43 - 56, Total Non-Gushing | 25
  Participant 1, F Day 57 - 70 , Total Gushing | 4
  Participant 1, F Day 57 - 70 , Total Non-Gushing | 17
  Participant 1, F Day 71 - 84 , Total Gushing | 0
  Participant 1, F Day 71 - 84 , Total Non-Gushing | 23
  Participant 1, F Day 85 - 98 , Total Gushing | 4
  Participant 1, F Day 85 - 98 , Total Non-Gushing | 27
  Participant 1, F Day 99 - 112 , Total Gushing | 6
  Participant 1, F Day 99 - 112 , Total Non-Gushing | 28
  Participant 2, Baseline, Total Gushing | 25
  Participant 2, Baseline, Total Non-Gushing | 17
  Participant 2, OT Day1-5, Total Gushing | 5
  Participant 2, OT Day1-5, Total Non-Gushing | 12
  Participant 2, OT Day 6 - 19 , Total Gushing | 24
  Participant 2, OT Day 6 - 19 , Total Non-Gushing | 18
  Participant 2, OT Day 20 - 33 , Total Gushing | 17
  Participant 2, OT Day 20 - 33 , Total Non-Gushing | 38
  Participant 2, OT Day 34 - 47, Total Gushing | 10
  Participant 2, OT Day 34 - 47 , Total Non-Gushing | 34
  Participant 2, OT Day 48 - 61 , Total Gushing | 10
  Participant 2, OT Day 48 - 61 , Total Non-Gushing | 22
  Participant 2, OT Day 62 - 75 , Total Gushing | 20
  Participant 2, OT Day 62 - 75 , Total Non-Gushing | 22
  Participant 2, OT Day 76 - 89 , Total Gushing | 17
  Participant 2, OT Day 76 - 89 , Total Non-Gushing | 20
  Participant 2, F Day 1 - 14 , Total Gushing | 14
  Participant 2, F Day 1 - 14 , Total Non-Gushing | 18
  Participant 2, F Day 15 - 28 , Total Gushing | 14
  Participant 2, F Day 15 - 28 , Total Non-Gushing | 7
  Participant 2, F Day 29 - 42 , Total Gushing | 18
  Participant 2, F Day 29 - 42 , Total Non-Gushing | 10
  Participant 2, F Day 43 - 56 , Total Gushing | 17
  Participant 2, F Day 43 - 56 , Total Non-Gushing | 11
  Participant 2, F Day 57 - 70 , Total Gushing | 14
  Participant 2, F Day 57 - 70 , Total Non-Gushing | 19
  Participant 2, F Day 71 - 84 , Total Gushing | 9
  Participant 2, F Day 71 - 84 , Total Non-Gushing | 19
  Participant 2, F Day 85 - 98 , Total Gushing | 13
  Participant 2, F Day 85 - 98 , Total Non-Gushing | 21
  Participant 2, F Day 99 , Total Gushing | 1
  Participant 2, F Day 99, Total Non-Gushing | 2
  Participant 3, Baseline , Total Gushing | 10
  Participant 3, Baseline, Total Non-Gushing | 1
  Participant 3, OT Day1 - 14 , Total Gushing | 8
  Participant 3, OT Day1 - 14 , Total Non-Gushing | 9
  Participant 3, OT Day 15 - 28 , Total Gushing | 7
  Participant 3, OT Day 15 - 28 , Total Non-Gushing | 9
  Participant 3, OT Day 29 - 42 , Total Gushing | 12
  Participant 3, OT Day 29 - 42 , Total Non-Gushing | 1
  Participant 3, OT Day 43 - 56 , Total Gushing | 6
  Participant 3, OT Day 43 - 56 , Total Non-Gushing | 5
  Participant 3, OT Day 57 - 70 , Total Gushing | 4
  Participant 3, OT Day 57 - 70 , Total Non-Gushing | 4
  Participant 3, OT Day 71 - 84 , Total Gushing | 7
  Participant 3, OT Day 71 - 84 , Total Non-Gushing | 6
  Participant , F Day 1 - 14 , Total Gushing | 9
  Participant , F Day 1 - 14 , Total Non-Gushing | 3
  Participant 3, F Day 15 - 28 , Total Gushing | 0
  Participant 3, F Day 15 - 28 , Total Non-Gushing | 3
  Participant 3, F Day 29 - 42, Total Gushing | 4
  Participant 3, F Day 29 - 42 , Total Non-Gushing | 4
  Participant 3, F Day 43 - 56 , Total Gushing | 7
  Participant 3, F Day 43 - 56 , Total Non-Gushing | 4
  Participant 3, F Day 57 - 70 , Total Gushing | 6
  Participant 3, F Day 57 - 70 , Total Non-Gushing | 5
  Participant 3, F Day 71 - 84 , Total Gushing | 4
  Participant 3, F Day 71 - 84 , Total Non-Gushing | 1
  Participant 3, F Day 85 - 98 , Total Gushing | 4
  Participant 3, F Day 85 - 98 , Total Non-Gushing | 1
  Participant 3, F Day 99 - 112 , Total Gushing | 6
  Participant 3, F Day 99 - 112 , Total Non-Gushing | 3
  Participant 3, F Day 113 - 115 , Total Gushing | 0
  Participant 3, F Day 113 - 115 , Total Non-Gushing | 2
  Participant 4, Baseline, Total Gushing | 3
  Participant 4, Baseline, Total Non-Gushing | 24
  Participant 4, OT Day1, Total Gushing | 1
  Participant 4, OT Day1, Total Non-Gushing | 0
  Participant 4, OT Day 2 - 15 , Total Gushing | 9
  Participant 4, OT Day 2 - 15 , Total Non-Gushing | 19
  Participant 4, OT Day 16 - 29 , Total Gushing | 2
  Participant 4, OT Day 16 - 29 , Total Non-Gushing | 16
  Participant 4, OT Day 30 - 43 , Total Gushing | 2
  Participant 4, OT Day 30 - 43 , Total Non-Gushing | 17
  Participant 4, OT Day 44 - 57 , Total Gushing | 2
  Participant 4, OT Day 44 - 57 , Total Non-Gushing | 15
  Participant 4, OT Day 58 - 71 , Total Gushing | 1
  Participant 4, OT Day 58 - 71 , Total Non-Gushing | 6
  Participant 4, OT Day 72 - 85 , Total Gushing | 0
  Participant 4, OT Day 72 - 85 , Total Non-Gushing | 6
  Participant 4, F Day 1-14, Total Gushing | 0
  Participant 4, F Day 1-14, Total Non-Gushing | 6
  Participant 4, F Day 15 - 28 , Total Gushing | 0
  Participant 4, F Day 15 - 28 , Total Non-Gushing | 9
  Participant 4, F Day 29 - 42 , Total Gushing | 6
  Participant 4, F Day 29 - 42 , Total Non-Gushing | 12
  Participant 4, F Day 43 - 56 , Total Gushing | 2
  Participant 4, F Day 43 - 56 , Total Non-Gushing | 10
  Participant 4, F Day 57 - 70 , Total Gushing | 3
  Participant 4, F Day 57 - 70 , Total Non-Gushing | 16
  Participant 4, F Day 71 - 84 , Total Gushing | 0
  Participant 4, F Day 71 - 84 , Total Non-Gushing | 11
  Participant 4, F Day 85 - 98 , Total Gushing | 3
  Participant 4, F Day 85 - 98 , Total Non-Gushing | 9
  Participant 4, F Day 99 - 112 , Total Gushing | 3
  Participant 4, F Day 99 - 112 , Total Non-Gushing | 11
  Participant 4, F Day 113 - 120 , Total Gushing | 2
  Participant 4, F Day 113 - 120 , Total Non-Gushing | 8
  Participant 5, Baseline, Total Gushing | 13
  Participant 5, Baseline, Total Non-Gushing | 22
  Participant 5, OT Day 1 - 2 , Total Gushing | 2
  Participant 5, OT Day 1 - 2 , Total Non-Gushing | 4
  Participant 5 OT Day 3 - 16 , Total Gushing | 11
  Participant 5 OT Day 3 - 16 , Total Non-Gushing | 22
  Participant 5, OT Day 17 - 30 , Total Gushing | 15
  Participant 5, OT Day 17 - 30 , Total Non-Gushing | 22
  Participant 5, OT Day 31 - 44 , Total Gushing | 11
  Participant 5, OT Day 31 - 44 , Total Non-Gushing | 23
  Participant 5, OT Day 45 - 58 , Total Gushing | 4
  Participant 5, OT Day 45 - 58 , Total Non-Gushing | 24
  Participant 5, OT Day 59 - 72 , Total Gushing | 6
  Participant 5, OT Day 59 - 72 , Total Non-Gushing | 28
  Participant 5, OT Day 73 - 86, Total Gushing | 4
  Participant 5, OT Day 73 - 86 , Total Non-Gushing | 26
  Participant 5, F Day 1-14, Total Gushing | 3
  Participant 5, F Day 1-14, Total Non-Gushing | 27
  Participant 5, F Day 15 - 28 , Total Gushing | 4
  Participant 5, F Day 15 - 28 , Total Non-Gushing | 15
  Participant 5, F Day 29 - 42, Total Gushing | 12
  Participant 5, F Day 29 - 42 , Total Non-Gushing | 10
  Participant 5, F Day 43 - 56 , Total Gushing | 6
  Participant 5, F Day 43 - 56 , Total Non-Gushing | 17
  Participant 5, F Day 57 - 70 , Total Gushing | 13
  Participant 5, F Day 57 - 70 , Total Non-Gushing | 15
  Participant 5, F Day 71 - 84 , Total Gushing | 9
  Participant 5, F Day 71 - 84 , Total Non-Gushing | 16
  Participant 5, F Day 85 - 98 , Total Gushing | 11
  Participant 5, F Day 85 - 98 , Total Non-Gushing | 16
  Participant 5, F Day 99 - 112 , Total Gushing | 13
  Participant 5, F Day 99 - 112 , Total Non-Gushing | 18
  Participant 5, F Day 113 - 118 , Total Gushing | 5
  Participant 5, F Day 113 - 118 , Total Non-Gushing | 4
  Participant 6, Baseline, Total Gushing | 0
  Participant 6, Baseline, Total Non-Gushing | 18
  Participant 6, OT Day 1, Total Gushing | 0
  Participant 6, OT Day 1 , Total Non-Gushing | 0
  Participant 6, OT Day 2 - 15 , Total Gushing | 0
  Participant 6, OT Day 2 - 15 , Total Non-Gushing | 13
  Participant 6, OT Day 16 - 29 , Total Gushing | 0
  Participant 6, OT Day 16 - 29 , Total Non-Gushing | 28
  Participant 6, OT Day 30 - 43 , Total Gushing | 0
  Participant 6, OT Day 30 - 43 , Total Non-Gushing | 19
  Participant 6, F Day 1-14, Total Gushing | 0
  Participant 6, F Day 1-14, Total Non-Gushing | 17
  Participant 6, F Day 15 - 28 , Total Gushing | 0
  Participant 6, F Day 15 - 28 , Total Non-Gushing | 13
  Participant 6, F Day 29 - 42 , Total Gushing | 0
  Participant 6, F Day 29 - 42 , Total Non-Gushing | 9
  Participant 6, F Day 43 - 56 , Total Gushing | 0
  Participant 6, F Day 43 - 56 , Total Non-Gushing | 17
  Participant 7, Baseline, Total Gushing | 3
  Participant 7, Baseline, Total Non-Gushing | 10
  Participant 7, OT Day 1 - 14 , Total Gushing | 3
  Participant 7, OT Day 1 - 14 , Total Non-Gushing | 6
  Participant 7, OT Day 15 - 28 , Total Gushing | 0
  Participant 7, OT Day 15 - 28 , Total Non-Gushing | 5
  Participant 7, OT Day 29 - 42 , Total Gushing | 2
  Participant 7, OT Day 29 - 42 , Total Non-Gushing | 9
  Participant 7, OT Day 43 - 56 , Total Gushing | 2
  Participant 7, OT Day 43 - 56 , Total Non-Gushing | 3
  Participant 7, OT Day 57 - 70 , Total Gushing | 1
  Participant 7, OT Day 57 - 70 , Total Non-Gushing | 4
  Participant 7, OT Day 71 - 84 , Total Gushing | 3
  Participant 7, OT Day 71 - 84 , Total Non-Gushing | 3
  Participant 7, F Day 1-14, Total Gushing | 2
  Participant 7, F Day 1-14, Total Non-Gushing | 5
  Participant 7, F Day 15 - 28 , Total Gushing | 6
  Participant 7, F Day 15 - 28 , Total Non-Gushing | 6
  Participant 7, F Day 29 - 42 , Total Gushing | 3
  Participant 7, F Day 29 - 42 , Total Non-Gushing | 4
  Participant 7, F Day 43 - 54 , Total Gushing | 3
  Participant 7, F Day 43 - 54 , Total Non-Gushing | 3

7. Primary Outcome: Total Iron Intake Over the Last 4 Weeks of the Dosing Period
Description: Total iron intake at Baseline is defined as the sum total of iron intake (oral + intravenous infusion) during the last 4 weeks of run-in period (i.e., Day -28 to Day -1). Total iron intake over the last 4 weeks of run-in and during last 4 weeks of dosing period was listed. Individual participant data has been reported.
Time Frame: Last 4 weeks of run-in and during last 4 weeks of dosing period
Population: Pharmacodynamic Population
Measure: Number; unit: Milligram
Arm/Group | GW786034 50 mg Once Daily
Number analyzed (Participants) | 7
Milligram
  Participant 1, Baseline | 300
  Participant 1, Dosing period, Day 1 - 27 | 300
  Participant 1, Dosing period, Day 28 - 55 | 300
  Participant 1, Dosing period, Day 56 - 83 | 600
  Participant 2, Baseline | 1000
  Participant 2, Dosing period, Day 1 - 5 | 0
  Participant 2, Dosing period, Day 6 - 33 | 2000
  Participant 2, Dosing period, Day 34 - 61 | 1000
  Participant 2, Dosing period, Day 62 - 89 | 1000
  Participant 3, Baseline | 3000
  Participant 3, Dosing period, Day 1 - 28 | 1000
  Participant 3, Dosing period, Day 29 - 56 | 1000
  Participant 3, Dosing period, Day 57 - 84 | 2000
  Participant 4, Baseline | 800
  Participant 4, Dosing period, Day 1 | 0
  Participant 4, Dosing period, Day 2 - 29 | 800
  Participant 4, Dosing period, Day 30 - 57 | 400
  Participant 4, Dosing period, Day 58 - 85 | 300
  Participant 5, Baseline | 750
  Participant 5, Dosing period, Day 1 - 2 | 0
  Participant 5, Dosing period, Day 3 - 30 | 0
  Participant 5, Dosing period, Day 31 - 58 | 1500
  Participant 5, Dosing period, Day 59 - 86 | 0
  Participant 6, Baseline | 4150
  Participant 6, Dosing period, Day 1 - 15 | 2460
  Participant 6, Dosing period, Day 16 - 43 | 3640
  Participant 7, Baseline | 510
  Participant 7, Dosing period, Day 1 - 28 | 510
  Participant 7, Dosing period, Day 29 - 56 | 0
  Participant 7, Dosing period, Day 57 - 84 | 1020

8. Primary Outcome: Total Iron Intake Over the Entire Dosing and Follow-up Period by 4 Week Interval
Description: Total iron intake at Baseline is defined as the sum total of iron intake (oral + intravenous infusion) during the last 4 weeks of run-in period (i.e., Day -28 to Day -1). Total iron intake over the entire dosing and follow-up period was listed by 4 week interval. Individual participant data has been reported.
Time Frame: Last 4 weeks of run-in and during last 4 weeks of dosing period
Population: Pharmacodynamic Population
Measure: Number; unit: Milligram
Arm/Group | GW786034 50 mg Once Daily
Number analyzed (Participants) | 7
Milligram
  Participant 1, Baseline | 300
  Participant 1, Dosing period, Day 1 - 27 | 300
  Participant 1, Dosing period, Day 28 - 55 | 300
  Participant 1, Dosing period, Day 56 - 83 | 600
  Participant 1, Follow up, Day 1 - 28 | 0
  Participant 1, Follow up, Day 29 - 56 | 300
  Participant 1, Follow up, Day 57 - 84 | 600
  Participant 1, Follow up, Day 85 - 112 | 0
  Participant 2, Baseline | 1000
  Participant 2, Dosing period, Day 1 - 5 | 0
  Participant 2, Dosing period, Day 6 - 33 | 2000
  Participant 2, Dosing period, Day 34 - 61 | 1000
  Participant 2, Dosing period, Day 62 - 89 | 1000
  Participant 2, Follow up, Day 1 - 28 | 1000
  Participant 2, Follow up, Day 29 - 56 | 500
  Participant 2, Follow up, Day 57 - 84 | 1500
  Participant 2, Follow up, Day 85 - 106 | 500
  Participant 3, Baseline | 3000
  Dosing period, Day 1 - 28 | 1000
  Participant 3, Dosing period, Day 29 - 56 | 1000
  Participant 3, Dosing period, Day 57 - 84 | 2000
  Participant 3, Follow up, Day 1 - 28 | 3000
  Participant 3, Follow up, Day 29 - 56 | 1000
  Participant 3, Follow up, Day 57 - 84 | 2000
  Participant 3, Follow up, Day 85 - 112 | 2000
  Participant 3, Follow up, Day 113 | 1000
  Participant 4, Baseline | 800
  Participant 4, Dosing period, Day 1 | 0
  Participant 4, Dosing period, Day 2 - 29 | 800
  Participant 4, Dosing period, Day 30 - 57 | 400
  Participant 4, Dosing period, Day 58 - 85 | 300
  Participant 4, Follow up, Day 1 - 28 | 100
  Participant 4, Follow up, Day 29 - 56 | 200
  Participant 4, Follow up, Day 57 - 84 | 200
  Participant 4, Follow up, Day 85 - 112 | 200
  Participant 4, Follow up, Day 113 | 0
  Participant 5, Baseline | 750
  Participant 5, Dosing period, Day 1 - 2 | 0
  Participant 5, Dosing period, Day 3 - 30 | 0
  Participant 5, Dosing period, Day 31 - 58 | 1500
  Participant 5, Dosing period, Day 59 - 86 | 0
  Participant 5, Follow up, Day 1 - 28 | 0
  Participant 5, Follow up, Day 29 - 56 | 750
  Participant 5, Follow up, Day 57 - 84 | 0
  Participant 5, Follow up, Day 85 - 112 | 750
  Participant 5, Follow up, Day 113 | 0
  Participant 6, Baseline | 4150
  Participant 6, Dosing period, Day 1 - 15 | 2460
  Participant 6, Dosing period, Day 16 - 43 | 3640
  Participant 6, Follow up, Day 1 - 28 | 3640
  Participant 6, Follow up, Day 29 - 56 | 4660
  Participant 7, Baseline | 510
  Participant 7, Dosing period, Day 1 - 28 | 510
  Participant 7, Dosing period, Day 29 - 56 | 0
  Dosing period, Day 57 - 84 | 1020
  Participant 7, Follow up, Day 1 - 28 | 0
  Participant 7, Follow up, Day 29 - 55 | 1020

9. Primary Outcome: Total Units of Packed Red Blood Cells (PRBCs) Transfused During the Entire Dosing and Follow-up Period by 4 Week Interval
Description: Baseline PRBC transfused is defined as the number of units of PRBC transfused during the last 4 weeks of run-in period (i.e., Day -28 to Day -1). Total units of PRBCs transfused during the entire dosing and follow-up period was listed by 4 week interval. Individual participant data been reported.
Time Frame: Over the last 4 weeks of run-in and at 4 week intervals during dosing and follow-up
Population: Pharmacodynamic Population
Measure: Number; unit: Number of units
Arm/Group | GW786034 50 mg Once Daily
Number analyzed (Participants) | 7
Number of units
  Participant 1, Baseline | 0
  Participant 1, Dosing period, Day 1 - 27 | 0
  Participant 1, Dosing period, Day 28 - 55 | 0
  Participant 1, Dosing period, Day 56 - 83 | 0
  Participant 1, Follow up, Day 1 - 28 | 0
  Participant 1, Follow up, Day 29 - 56 | 0
  Participant 1, Follow up, Day 57 - 84 | 0
  Participant 1, Follow up, Day 85 - 112 | 0
  Participant 2, Baseline | 0
  Participant 2, Dosing period, Day 1 - 5 | 0
  Participant 2, Dosing period, Day 6 - 33 | 0
  Participant 2, Dosing period, Day 34 - 61 | 0
  Participant 2, Dosing period, Day 62 - 89 | 0
  Participant 2, Follow up, Day 1 - 28 | 0
  Participant 2, Follow up, Day 29 - 56 | 0
  Participant 2, Follow up, Day 57 - 84 | 0
  Participant 2, Follow up, Day 85 - 106 | 0
  Participant 3, Baseline | 2
  Participant 3, Dosing period, Day 1 - 28 | 2
  Participant 3, Dosing period, Day 29 - 56 | 0
  Participant 3, Dosing period, Day 57 - 84 | 0
  Participant 3, Follow up, Day 1 - 28 | 0
  Participant 3, Follow up, Day 29 - 56 | 0
  Participant 3, Follow up, Day 57 - 84 | 0
  Participant 3, Follow up, Day 85 - 112 | 2
  Participant 3, Follow up, Day 113 | 0
  Participant 4, Baseline | 0
  Participant 4, Dosing period, Day 1 | 0
  Participant 4, Dosing period, Day 2 - 29 | 0
  Participant 4, Dosing period, Day 30 - 57 | 0
  Participant 4, Dosing period, Day 58 - 85 | 0
  Participant 4, Follow up, Day 1 - 28 | 0
  Participant 4, Follow up, Day 29 - 56 | 0
  Participant 4, Follow up, Day 57 - 84 | 0
  Participant 4, Follow up, Day 85 - 112 | 0
  Participant 4, Follow up, Day 113 | 0
  Participant 5, Baseline | 0
  Participant 5, Dosing period, Day 1 - 2 | 0
  Participant 5, Dosing period, Day 3 - 30 | 0
  Participant 5, Dosing period, Day 31 - 58 | 0
  Participant 5, Dosing period, Day 59 - 86 | 0
  Participant 5, Follow up, Day 1 - 28 | 0
  Participant 5, Follow up, Day 29 - 56 | 0
  Participant 5, Follow up, Day 57 - 84 | 0
  Participant 5, Follow up, Day 85 - 112 | 2
  Participant 5, Follow up, Day 113 | 0
  Participant 6, Baseline | 0
  Participant 6, Dosing period, Day 1 - 15 | 0
  Participant 6, Dosing period, Day 16 - 43 | 0
  Participant 6, Follow up, Day 1 - 28 | 0
  Participant 6, Follow up, Day 29 - 56 | 0
  Participant 7, Baseline | 0
  Participant 7, Dosing period, Day 1 - 28 | 0
  Participant 7, Dosing period, Day 29 - 56 | 0
  Participant 7, Dosing period, Day 57 - 84 | 0
  Participant 7, Follow up, Day 1 - 28 | 0
  Participant 7, Follow up, Day 29 - 55 | 0

10. Secondary Outcome: Change From Baseline in the Average of the Last 3 Ferritin Measures in the Dosing Period (Week 9, Week 10.5 and Week 12)
Description: For post-Baseline ferritin assessments, average of the last 3 measurements of the dosing period (Weeks 9, 10.5 and 12) was computed. Only pre-infusion ferritin values have been included in the analyses. Baseline ferritin value is the average of the last two measurements during the run-in period. Average of the last two measurements during the run-in period was calculated as sum of the last 2 measured values of ferritin divided by 2. Change from Baseline was calculated as the average of the last 3 measured values of ferritin minus the Baseline value. Average of the last 3 measurements was calculated as sum of the last 3 measured values of ferritin divided by 3. If measurements were missing at one or two of the 3 visits at Weeks 9, 10.5 and 12, then the average was based on the available measurements.
Time Frame: Baseline, Week 9, Week 10.5 and Week 12
Population: Pharmacodynamic Population. Only those par. available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: micrograms per liter (µg per L)
Arm/Group | GW786034 50 mg Once Daily
Number analyzed (Participants) | 6
micrograms per liter (µg per L) | -73.17 (115.016)

11. Secondary Outcome: Change From Baseline in Ferritin at the Indicated Time Points
Description: Only pre-infusion ferritin values have been included in the analyses. All ferritin measurements that fall within 5 days of iron infusion date are considered post-infusion. Baseline ferritin value is defined as the average of the last two measurements during the run-in period. Average of the last two measurements during the run-in period was calculated as sum of the last 2 measured values of ferritin divided by 2. Change from Baseline is calculated as the difference between the Post dose value at indicated visit minus Baseline value. Par. were evaluated at baseline, treatment period (Weeks 1.5, 3, 4.5, 6, 7.5, 9, 10.5 and 12) and follow-up period (16, 20, 24 and 28).
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: µg per L
Arm/Group | GW786034 50 mg Once Daily
Number analyzed (Participants) | 7
µg per L
  Week 1.5, n=4 | -73.75 (223.827)
  Week 3, n=6 | -59.33 (182.538)
  Week 4.5, n=5 | -118.30 (184.946)
  Week 6, n=7 | 7.07 (62.727)
  Week 7.5, n=2 | -31.75 (67.529)
  Week 9, n=6 | -48.83 (86.762)
  Week 10.5, n=5 | -82.90 (127.769)
  Week 12, n=3 | -111.67 (231.107)
  Follow-Up Week 16, n=7 | -85.36 (154.078)
  Follow-Up Week 20, n=6 | -14.56 (119.056)
  Follow-Up Week 24, n=4 | -70.25 (237.869)
  Follow-Up Week 28, n=5 | 1.90 (82.750)

12. Secondary Outcome: Overall Health-related (HR) Quality of Life (QOL) Score Measured Using SF-36v2 at Day 1, Week 6 and Week 12
Description: SF-36v2 is a generic HR QOL instrument with 36 items covering 8 subscales (SS) clustering into 2 global scores, the physical component summary score (PCS: physical functioning (PF), role physical (RP), bodily pain (BP), and general health (GH)) and mental component summary score (MCS: vitality (VT), social functioning (SF), role emotional (RE) and mental health (MH)). All scores are normalized so that mean score for a representative US population = 50, with a standard deviation = 10. Information was used to observe a direction in overall QOL. Ranges are shown below. Higher scores represent better QOL and minimum important differences are PF, 3; RP, 3; BP, 3; GH, 2; VT, 2; SF, 3; RE, 4; and MH, 3 PCS, 2; MCS, 3. Response Consistency Index (RCI) measures the consistency of responses to individual survey responses. Lower the score the more consistent the individual responses. SF-6D Health Utility Index (HUI) Score = 0 (worst measured health state) to 1 (best measured health state).
Time Frame: Day (D) 1, Week (W) 6 and Week 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | GW786034 50 mg Once Daily
Number analyzed (Participants) | 7
Scores on a scale
  BP (0-100 score), D1, n=7 | 58.29 (20.966)
  BP (0-100 score), W6, n=7 | 70.86 (29.396)
  BP (0-100 score), W12, n=6 | 53.67 (19.232)
  GH (0-100 score), D1, n=7 | 50.14 (28.510)
  GH (0-100 score), W6, n=7 | 51.86 (26.448)
  GH (0-100 score), W12, n=6 | 49.67 (17.351)
  MH (0-100 score), D1, n=7 | 61.43 (22.678)
  MH (0-100 score), W6, n=7 | 70.00 (21.602)
  MH (0-100 score), W12, n=6 | 71.67 (12.111)
  PF (0-100 score), D1, n=7 | 52.86 (26.590)
  PF (0-100 score), W6, n=7 | 55.72 (24.397)
  PF (0-100 score), W12, n=6 | 68.33 (12.906)
  RE (0-100 score), D1, n=7 | 63.10 (31.861)
  RE (0-100 score), W6, n=7 | 83.33 (23.570)
  RE (0-100 score), W12, n=6 | 75.00 (16.667)
  RP (0-100 score), D1, n=7 | 58.04 (30.129)
  RP (0-100 score), W6, n=7 | 66.96 (23.583)
  RP (0-100 score), W12, n=6 | 66.67 (25.820)
  SF (0-100 score), D1, n=7 | 66.07 (25.733)
  SF (0-100 score), W6, n=7 | 83.93 (17.252)
  SF (0-100 score), W12, n=6 | 62.50 (20.917)
  VT (0-100 score), D1, n=7 | 42.86 (18.196)
  VT (0-100 score), W6, n=7 | 53.57 (20.684)
  VT (0-100 score), W12, n=6 | 47.92 (11.637)
  BP(norm-based score), D1, n=7 (21.68-62.0 score) | 44.40 (8.278)
  BP(norm-based score), W6, n=7 (21.68-62.0 score) | 49.37 (11.605)
  BP(norm-based score), W12, n=6 (21.68-62.0 score) | 42.58 (7.592)
  GH(norm-based score), D1, n=7 (18.95-66.5 score) | 43.41 (12.577)
  GH(norm-based score), W6, n=7 (18.95-66.5 score) | 44.17 (11.666)
  GH(norm-based score), W12, n=6 (18.95-66.5 score) | 43.20 (7.655)
  MH(norm-based score), D1, n=7 (11.63-63.95 score) | 43.56 (11.237)
  MH(norm-based score), W6, n=7 (11.63-63.95 score) | 47.81 (10.704)
  MH(norm-based score), W12, n=6 (11.63-63.95 score) | 48.63 (6.002)
  PF(norm-based score), D1, n=7 (19.26-57.54 score) | 39.41 (10.256)
  PF(norm-based score), W6, n=7 (19.26-57.54 score) | 40.52 (9.410)
  PF(norm-based score),W12, n=6 (19.26-57.54 score) | 45.38 (4.979)
  RE(norm-based score), D1, n=7 (14.39-56.17 score) | 38.74 (14.593)
  RE(norm-based score), W6, n=7 (14.39-56.17 score) | 48.01 (10.795)
  RE(norm-based score), W12, n=6 (14.39-56.17 score) | 44.19 (7.635)
  RP(norm-based score), D1, n=7 (21.23-57.16 score) | 42.34 (10.614)
  RP(norm-based score), W6, n=7 (21.23-57.16 score) | 45.48 (8.308)
  RP(norm-based score), W12, n=6 (21.23-57.16 score) | 45.38 (9.096)
  SF(norm-based score), D1, n=7 (17.23-57.34 score) | 50.38 (6.823)
  SF(norm-based score), W6, n=7 (17.23-57.34 score) | 43.32 (10.174)
  SF(norm-based score), W12,n=6 (17.23-57.34 score) | 41.91 (8.270)
  VT(norm-based score), D1, n=7 (22.89-70.4 score) | 44.26 (7.923)
  VT(norm-based score), W6, n=7 (22.89-70.4 score) | 48.93 (9.007)
  VT(norm-based score), W12, n=6 (22.89-70.4 score) | 46.47 (5.069)
  PCS, D1, n=7 (5.02-79.78 score) | 42.87 (7.767)
  PCS, W6, n=7 (5.02-79.78 score) | 43.57 (9.507)
  PCS, W12, n=6 (5.02-79.78 score) | 43.74 (6.743)
  MCS, D1, n=7 (-3.33-80.09 score) | 42.87 (12.198)
  MCS, W6, n=7 (-3.33-80.09 score) | 50.81 (9.652)
  MCS, W12, n=6 (-3.33-80.09 score) | 46.27 (6.933)
  RCI, D1, n=7 (0-15 score) | 0.00 (0.000)
  RCI, W6, n=7 (0-15 score) | 0.00 (0.000)
  RCI, W12, n=6 (0-15 score) | 0.00 (0.000)
  SF-6D HUI Score, D1, n=7 (0-1 score) | 0.64 (0.114)
  SF-6D HUI Score, W6, n=7 (0-1 score) | 0.70 (0.114)
  SF-6D HUI Score, W12, n=6 (0-1 score) | 0.64 (0.051)
  MH Enhanced Score, D1, n=7 (0-63 score) | 11.57 (7.955)
  MH Enhanced Score, W6, n=7 (0-63 score) | 8.62 (7.459)
  MH Enhanced Score, W12, n=6 (0-63 score) | 7.83 (3.939)

13. Secondary Outcome: Number of Participants With the Indicated Clinical Chemistry Values of Potential Clinical Concern
Description: The following laboratory parameters were analyzed: hemoglobin, hematocrit, red blood cell count, platelet count, white blood cell count, total neutrophils, lymphocytes; alanine amino transferase (ALT), alkaline phosphatase (ALP), aspartate amino transferase (AST), gamma glutamyl transferase (GGT), total bilirubin, albumin, total protein, blood urea nitrogen, creatinine, uric acid, sodium, potassium, chloride, calcium, total carbondioxide, glucose, magnesium, and ferritin. Only those parameters for which at least one value of clinical concern are reported in the table. Values above upper limit of normal and below lower limit to normal have been presented as high and low respectively.
Time Frame: Up to Week 16
Population: Safety Population: The Safety Population comprises of all participants who received at least one dose of study treatment. This population is based on the treatment the participant actually received.
Measure: Number; unit: Participants
Arm/Group | GW786034 50 mg Once Daily
Number analyzed (Participants) | 7
Participants
  ALP, High | 1
  ALP, Low | 0
  ALT, High | 1
  ALT, Low | 0
  AST, High | 1
  AST, Low | 0
  Calcium, High | 0
  Calcium, Low | 1
  Ferritin, High | 0
  Ferrtin, Low | 4
  GGT, High | 3
  GGT, Low | 0
  Glucose, High | 0
  Glucose, Low | 3
  Hemoglobin, High | 0
  Hemoglobin, Low | 4
  Hematocrit, High | 0
  Hematocrit, Low | 2
  Lymphocytes, High | 0
  Lymphocytes, Low | 1
  Platelet count, High | 1
  Platelet count, Low | 0
  Total Protein, High | 0
  Total Protein, Low | 1
  WBC, High | 0
  WBC, Low | 3

14. Secondary Outcome: Number of Participants With Vital Signs Data Meeting Criteria of Potential Clinical Concern
Description: The following laboratory parameters were analyzed in supine position after 10 minutes rest: Diastolic blood pressure (DBP), Systolic blood pressure (SBP) and Heart rate (HR). Values above upper limit of normal and below lower limit to normal have been presented as high and low respectively.
Time Frame: Up to Week 16
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | GW786034 50 mg Once Daily
Number analyzed (Participants) | 7
Participants
  DBP, Anytime OT, High,n=7 | 0
  DBP, Anytime OT, Low, n=7 | 1
  DBP, Day 1, High, n=7 | 0
  DBP, Day 1, Low, n=7 | 0
  DBP, Week 3, High, n=7 | 0
  DBP, Week 3, Low, n=7 | 1
  DBP, Week 6, High, n=7 | 0
  DBP, Week 6, Low, n=7 | 0
  DBP, Week 9, High, n=6: number analyzed (Participants) | 6
  DBP, Week 9, High, n=6 | 0
  DBP, Week 9, Low, n=6: number analyzed (Participants) | 6
  DBP, Week 9, Low, n=6 | 0
  DBP, Week 12, High, n=6: number analyzed (Participants) | 6
  DBP, Week 12, High, n=6 | 0
  DBP, Week 12, Low, n=6: number analyzed (Participants) | 6
  DBP, Week 12, Low, n=6 | 0
  HR, Anytime OT, High, n=7 | 0
  HR, Anytime OT, Low, n=7 | 0
  HR, Day 1, High, n=7 | 0
  HR, Day 1, Low, n=7 | 0
  HR, Week 3, High, n=7 | 0
  HR, Week 3, Low, n=7 | 0
  HR, Week 6, High, n=7 | 0
  HR, Week 6, Low, n=7 | 0
  HR, Week 9, High, n=6: number analyzed (Participants) | 6
  HR, Week 9, High, n=6 | 0
  HR, Week 9, Low, n=6: number analyzed (Participants) | 6
  HR, Week 9, Low, n=6 | 0
  HR, Week 12, High, n=6: number analyzed (Participants) | 6
  HR, Week 12, High, n=6 | 0
  HR, Week 12, Low, n=6: number analyzed (Participants) | 6
  HR, Week 12, Low, n=6 | 0
  SBP, Anytime OT, High, n=7 | 0
  SBP, Anytime OT, Low, n=7 | 1
  SBP, Day 1, High, n=7 | 0
  SBP, Day 1, Low, n=7 | 1
  SBP, Week 3, High, n=7 | 0
  SBP, Week 3, Low, n=7 | 0
  SBP, Week 6, High, n=7 | 0
  SBP, Week 6, Low, n=7 | 0
  SBP, Week 9, High, n=6: number analyzed (Participants) | 6
  SBP, Week 9, High, n=6 | 0
  SBP, Week 9, Low, n=6: number analyzed (Participants) | 6
  SBP, Week 9, Low, n=6 | 0
  SBP, Week 12, High, n=6: number analyzed (Participants) | 6
  SBP, Week 12, High, n=6 | 0
  SBP, Week 12, Low, n=6: number analyzed (Participants) | 6
  SBP, Week 12, Low, n=6 | 0

15. Secondary Outcome: Number of Participants With Electrocardiogram (ECG) Data Meeting Criteria of Potential Clinical Concern
Description: The following ECG parameters were analyzed: PR, QRS, QT, corrected QT [QTc] intervals. Criteria for clinical concern:. QT where value is > 450, QT[QTc] where value is > 450, PR where value is < 110 or > 220, QRS where value is < 75 or >110.
Time Frame: Up to Week 16
Population: Safety population
Measure: Number; unit: Participants
Arm/Group | GW786034 50 mg Once Daily
Number analyzed (Participants) | 7
Participants | 1

16. Secondary Outcome: Number of Participants With Urinalysis Data Meeting Criteria of Potential Clinical Concern
Description: Protein - values of clinical concern if change from "trace" at baseline to 3+ any time on-therapy or from 0 at baseline to 2+ any time on-therapy.
Time Frame: Up to Week 16
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | GW786034 50 mg Once Daily
Number analyzed (Participants) | 7
Participants | 0

17. Secondary Outcome: Number of Participants With Any Adverse Events (AE) or Serious Adverse Event (SAE)
Description: An AE is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product.
Time Frame: From start of investigational product (IP) through the Study Phase (12 weeks post-dose) (assessed up to 28 weeks)
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | GW786034 50 mg Once Daily
Number analyzed (Participants) | 7
Participants
  Any AE | 7
  Serious AE | 0

18. Secondary Outcome: Plasma Concentration of GW786034 at the Indicated Time Points
Description: Predose (trough) blood samples were collected at weeks 3, 6, 9, and 12. Blood samples for pharmacokinetic (PK) profile were collected at pre-dose, 1, 2, 3, 4, 6 and 8 hours post dose. Area under the curve (0-tau), Concentration tau (Ctau), and maximum concentration (Cmax) following repeat administration was to be studied if data permitted.
Time Frame: Weeks 3, 6, 9 and 12
Population: Pharmacokinetic Population: The Pharmacokinetic Population includes participants who had a pharmacokinetic sample obtained and analyzed. Only those par. available at the indicated time points were analyzed (specified by n=X in the category titles).
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | GW786034 50 mg Once Daily
Number analyzed (Participants) | 7
µg/mL
  Week 3, n=7 | 6.3 (4.45)
  Week 6, n=7 | 6.5 (5.33)
  Week 9, n=6 | 6.2 (4.98)
  Week 12, n=6 | 6.8 (6.85)

19. Secondary Outcome: Graphical Exploration of PK/Pharmacodynamic (PD) Relationships Between Pazopanib Exposure and Selected PD
Description: Graphical exploration of PK/PD relationships between pazopanib exposure and selected parameters was to be explored if data permitted. Due to the small sample size and the fact that only one dose was studied these analyses were not performed.
Time Frame: Weeks 3, 6, 9 and 12
Population: Pharmacokinetic/Pharmacodynamic Population
Arm/Group | GW786034 50 mg Once Daily
Number analyzed (Participants) | 0

20. Secondary Outcome: PK/PD Modeling Analysis to Characterize the Relationship Between Pazopanib Trough Concentrations and Epistaxis Frequency and Duration/Severity
Description: A repeated categorical event per time interval PK/PD modeling analysis was planned (data permitting) to characterize the relationship between pazopanib trough concentrations and epistaxis frequency and duration/severity. Due to the small sample size and the fact that only one dose was studied these analyses were not performed.
Time Frame: Weeks 3, 6, 9 and 12
Population: Pharmacokinetic/Pharmacodynamic Population
Arm/Group | GW786034 50 mg Once Daily
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from start of IP through the Study Phase (12 weeks post-dose) to follow-up (assessed up to 28 weeks).
Description: On-treatment SAEs and non-serious AEs are reported for the Safety Population, which comprises of all randomized participants who received at least one dose of study treatment and is based on the actual study treatment received.
Arm/Group | GW786034 50 mg Once Daily
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 7/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GW786034 50 mg Once Daily (N=7)
Bronchitis (Infections and infestations) | 2
Nasopharyngitis (Infections and infestations) | 1
Otitis media (Infections and infestations) | 1
Pharyngitis streptococcal (Infections and infestations) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1
Alanine aminotransferase increased (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
Weight decreased (Investigations) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Muscle strain (Injury, poisoning and procedural complications) | 1
Sunburn (Injury, poisoning and procedural complications) | 1
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Confusional state (Psychiatric disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.